CLINICAL TRIAL: NCT00125138
Title: Safety and Efficacy of Melperone in the Treatment of Patients With Psychosis Associated With Parkinson's Disease
Brief Title: Melperone (an Anti-Psychotic) in Patients With Psychosis Associated With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lundbeck LLC (Industry)
Responsible Party: Lundbeck Inc., Lundbeck Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13104A; OV1003 (Other: Former study ID)
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-05

CONDITIONS: Parkinson's Disease; Psychotic Disorders
MeSH Terms: conditions — Parkinson Disease; Psychotic Disorders | interventions — metylperon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Melperone HCl - 20 mg (Experimental)
  Interventions: Drug: Melperone HCl
- Melperone HCl - 40 mg (Experimental)
  Interventions: Drug: Melperone HCl
- Melperone HCl - 60 mg (Experimental)
  Interventions: Drug: Melperone HCl
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melperone HCl — 20 mg/day. Strength of melperone syrup is 5 mg/mL
  Arms: Melperone HCl - 20 mg
Drug: Melperone HCl — 40 mg/day. Strength of melperone syrup is 5 mg/mL
  Arms: Melperone HCl - 40 mg
Drug: Melperone HCl — 60 mg/day. Strength of melperone syrup is 5 mg/mL
  Arms: Melperone HCl - 60 mg
Drug: Placebo — Syrup formulation
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of three target doses of melperone compared to placebo in the treatment of psychosis associated with Parkinson's disease. Subjects will be enrolled at approximately 20 investigational sites in the United States (U.S.) and 15 Ex-US sites. The maximum study duration will be 10 weeks. Subjects will have the option of continuing in an open-label extension study.

DETAILED DESCRIPTION:
Parkinson's Disease is a progressive neurodegenerative disorder characterized by bradykinesia, rigidity, tremor and abnormal posture and gait. Many patients can have mild to moderate symptoms, while others with advanced disease have symptoms which interfere with activities of daily living to a severe degree. Although effective in addressing motor dysfunction, long-term use of anti-Parkinsonian agents has been implicated as a component in the development of psychiatric side effects including psychosis. Treatment of psychosis with typical antipsychotics is not recommended in this patient population, since even low potency typical antipsychotics can cause marked exacerbations of parkinsonism in Parkinson's disease patients. The use of atypical antipsychotics (e.g., clozapine, risperidone and quetiapine) has shown some efficacy in the treatment of psychosis in PD patients. Melperone is classified atypical antipsychotic. European experience with melperone spans more than 30 years, and it encompasses an established antipsychotic efficacy profile in the treatment of confusion, anxiety, unrest (particularly in the elderly) and schizophrenia as well as a favorable safety and tolerability profile. Eligible subjects with Parkinson's disease psychosis will participate in a 1-2 week Screening/Washout Period, a 5 week Titration Phase (one of three doses of melperone or placebo), a 1 week Maintenance Phase and a Taper/Follow-up Period up to 2 weeks. Following the Day 43 assessment, subjects may be given the option of receiving melperone in an open-label extension study.

ELIGIBILITY:
Inclusion Criteria:

* The subject or subject's legally authorized representative (LAR) must sign and date the IRB/IEC approved Informed Consent Form and HIPAA Authorization (applicable to US sites only) prior to study participation.
* Male or female subjects. If female:

  * Subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or if of childbearing potential, must comply with a method of birth control acceptable to the investigator during the study, for at least one month prior to randomization and for one month following completion of the study.
  * Subject is not breastfeeding
  * Subjects of childbearing potential must have a negative serum pregnancy test at the screening visit and on Day 1.
* Subjects with a clinical diagnosis of idiopathic Parkinson's Disease, defined as the presence of at least three of the following cardinal features, in the absence of alternative explanations or atypical features:

  * Rest tremor
  * Rigidity
  * Bradykinesia and/or akinesia
  * Postural and gait abnormalities
* Subjects with psychosis:

  * Presence of visual and/or auditory hallucinations, with or without delusions, occurring during the four weeks prior to the screening visit.
  * Symptoms severe enough to clinically warrant treatment with an antipsychotic agent.
  * A Hallucinations or Delusions total item score (frequency x severity) of > 4 on the Neuropsychiatric Inventory (NPI).

    * Subjects currently being treated with an antipsychotic agent who have not had visual and/or auditory hallucinations, with or without delusions, during the four weeks prior to screening, and/or have a Hallucinations or Delusions total item score <4 on the NPI at the screening visit may be washed out (for 7 days or 5 half-lives, whichever is longer) and return for a repeat screening visit. The NPI Hallucinations or Delusions total item score must be ≥4 at the repeat visit to be considered for study entry.
* Subject is on a stable dose of anti-Parkinsonian medication(s) for at least 7 days or 5 half-lives, whichever is longer, prior to the screening visit and is expected to remain on a stable dose for the duration of the study.
* Subject is willing and able to comply with all study procedures.

Exclusion Criteria:

* Subject has any systemic factor contributing to the psychosis such as urinary infection, liver disease, renal failure, anemia, infection or cancer.
* Subject has a history of significant psychotic disorders prior to the diagnosis of Parkinson's Disease, including but not limited to schizophrenia or bipolar disorder.
* Subject has Dementia with Lewy-bodies (DLB).
* Subject has dementia or a major depressive disorder precluding accurate assessment on rating scales.
* Subject has an acute depressive episode at the time of the screening visit.
* A score on the Mini-Mental State Examination (MMSE) of < 21.
* Subject has had a dose adjustment of their antidepressant medication within 30 days prior to the screening visit, or dose adjustments are planned during the duration of the trial.
* Subject has had dose adjustments of an anxiolytic, cognitive enhancer, or other psychotropic medication (excluding antipsychotics) within 30 days prior to screening or dose adjustments are planned during the duration of the trial.
* Subject has received depot antipsychotic agents within the past 3 months.
* Subject has previously failed treatment with clozaril for psychosis in Parkinson's disease. Subjects who discontinued clozaril due to intolerability may be enrolled.
* Subject has used any investigational product within 30 days or 5 half-lives, whichever is longer, prior to screening.
* Subject cannot tolerate a wash-out of antipsychotic medication prior to randomization.
* Subject has a history of a serious respiratory, gastrointestinal, renal, hematologic or other medical disorder.
* Subject has a history of a serious cardiovascular condition (including, but not limited to, Class IV angina or Class IV heart failure) and/or a history of risk factors for Torsade de pointes (Tdp) (including but not limited to current treatment for hypokalemia or family history of long QT syndrome).
* Subject had myocardial infarction within 6 months prior to screening.
* Subject has a screening ECG with corrected QT interval by Bazett's correction formula (QTcB) of greater than 450 msec, if female, or 430 msec, if male.
* Subject requires treatment with an α-agonist agent.
* Subject has uncontrolled seizures, uncontrolled angina, or uncontrolled symptomatic orthostatic hypotension (or orthostatic hypotension leading to a history of falls 3 months prior to screening), or other medical disorders which would make the subject a poor candidate for a clinical trial.
* Subject has a history of severe adverse reactions to antipsychotic medications and/or quinine.
* Subject has clinically significant abnormal laboratory values, ECG, or findings on physical exam.
* Subject has a recent history or current evidence of substance dependence or abuse.
* Subject is unable to ingest liquid medication.
* Subject is currently being treated with Deep Brain Stimulation (DBS).

Randomization Criteria

* Subject has a Hallucinations or Delusions total item score (frequency x severity) of > 4 on the NPI.
* Female subjects of childbearing potential must have a negative serum pregnancy test.
* Subject has remained on a stable dose of anti-Parkinsonian medications.
* Subject has not had a dose adjustment in their antidepressant medication since the screening visit.
* Subjects have been washed out of previous antipsychotic agents for 5 half-lives or 7 days, whichever is longer, after the last dose of medication.
* Subject has not had dose adjustments in an anxiolytic, cognitive enhancer or other psychotropic medication (excluding antipsychotics) since the Screening Visit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-07; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (21):
- United States (10):
  - Northwest Neurospecialists, PLLC, Tucson, Arizona
  - Bradenton Research Center, Inc, Bradenton, Florida
  - University of South Florida, Tampa, Florida
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Quest Research Institute, Bingham Farms, Michigan
  - Struthers Parkinson's Center, Park Nicollet Health Services, Golden Valley, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Neurology Consultants of the Carolinas, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Neurology Associates, San Antonio, Texas
- India (8):
  - Department of Neurology, Rajendra Prasad Ward, King George Hospital, Visakhapatnam, Visakhapatnam, Andhra Pradesh
  - Department of Neurology, Manipal Hospital, Bangalore, Karnataka
  - M. S. Ramasah Memorial Hospital, Bangalore, Karnataka
  - KLE Hospital, Belgaum, Belagavi, Karnataka
  - Kasturra Medical College, Hospital, Attavar, Mangalore, Karnataka
  - SCTIMST, Trivandrum, Kerla
  - Jaslok Hospital and Research Center, Mumbai, Maharashtra
  - Apollo Hospitals Educational and Research Foundation, Chennai, Tamil Nadu
- Italy (3):
  - Fondazione Universita di Chieti C.E.S.I. Centro Studi sull'Invecchiamento, Chieti Scalo, Ambruzzo
  - U.O. Neurologia IRCCS San Raffaele Pisana, Rome, Lazio
  - IRCCS Centro Neurolesi "Bonino Pulejo", Messina, Sicily

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from July 2005 to December 2007. Investigator sites were hospitals, research centers, movement disorder centers, and neurology centers.
Pre-assignment Details: Subjects entered the Screening/Washout Period (for all previous antipsychotic medications) for a maximum of 2 weeks. On Day 1, the criteria for Randomization were reviewed by the investigator and psychiatric, motor function, and safety assessments were performed. Subjects who qualified on Day 1 were randomized to receive melperone or placebo.
Groups:
- Melperone HCl - 20 mg; Melperone HCl - 40 mg; Melperone HCl - 60 mg: 5 mg/mL Melperone syrup orally QHS
- Placebo: Syrup with 0.3 mg/mL quinine orally QHS
Period: Overall Study
Arm/Group | Melperone HCl - 20 mg | Melperone HCl - 40 mg | Melperone HCl - 60 mg | Placebo
Started | 15 | 20 (One subject requested withdrawal prior to treatment; data for the subject are excluded from results.) | 25 | 30
Completed | 12 | 17 | 21 | 25
Not Completed | 3 | 3 | 4 | 5
Not completed — Adverse Event | 1 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Sponsor decision-pt moved to assist care | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melperone HCl - 20 mg | Melperone HCl - 40 mg | Melperone HCl - 60 mg | Placebo | Total
Number analyzed (Participants) | 15 | 19 | 25 | 30 | 89
Age Continuous [Mean (Standard Deviation); unit: years] | 68.9 (6.2) | 69.0 (11.8) | 67.4 (11.2) | 68.5 (9.6) | 68.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10 | 10 | 30
  Male | 11 | 13 | 15 | 20 | 59

OUTCOME MEASURES:

1. Primary Outcome: Patient Evaluation of Symptoms of Psychosis.
Description: The change in the Scale for Assessment of Positive Symptoms (SAPS) total score. The SAPS total score ranges from 0 to 170, with higher scores indicating more severe psychosis.
Time Frame: 6 weeks (from Baseline to end of Maintenance Period)
Population: All randomized subjects who provided informed consent, took at least 1 dose of study drug, and had at least 1 post-baseline efficacy measurement (modified intent-to-treat [MITT] population) were included in the analysis of efficacy.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Melperone HCl - 20 mg | Melperone HCl - 40 mg | Melperone HCl - 60 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 21 | 25
Scores on a scale | -9.8 (4.4) | -12.9 (4.0) | -9.7 (3.5) | -10.0 (3.7)
Statistical Analysis 1: Comparison: Melperone HCl - 20 mg vs Placebo; The null hypothesis for each endpoint is that each melperone dose has the same mean as placebo; the alternative hypothesis is that at least one dose is more efficacious than placebo. Only subjects with both a baseline and Day 43 (end of Maintenance Phase) value are included; Test type: Superiority or Other; p = 0.5177, ANCOVA — One-sided pairwise p-value comparing each active treatment to placebo; One-way ANCOVA: Treatment, country, and baseline anti-psychotic medication status (recent or distant) as factors; baseline measurement as a covariate; Difference of LS Mean = 0.1, 95% CI 2-sided [-6.3 to 6.6]
Statistical Analysis 2: Comparison: Melperone HCl - 40 mg vs Placebo; The null hypothesis for each endpoint is that each melperone dose has the same mean as placebo; the alternative hypothesis hypothesis is that at least one dose is more efficacious than placebo. Only subjects with both a baseline and Day 43 (end of Maintenance Phase) value are included; Test type: Superiority or Other; p = 0.1519, ANCOVA — One-sided pairwise p-value comparing each active treatment to placebo; [statistical method as in outcome 1, analysis 1]; Difference of LS mean = -2.9, 95% CI 2-sided [-8.5 to 2.7]
Statistical Analysis 3: Comparison: Melperone HCl - 60 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5406, ANCOVA — One-sided pairwise p-value comparing each active treatment to placebo; [statistical method as in outcome 1, analysis 1]; Difference of LS mean = 0.3, 95% CI 2-sided [-5.2 to 5.8]

2. Secondary Outcome: Investigator/Caregiver Evaluations of Motor Function
Description: The change in the motor section of the Unified Parkinson's Disease Rating Scale (UPDRS III - motor exam) score. Scores on the UPDRS III - motor exam range from 0 to 108, with higher scores indicating more severe motor symptoms.
Time Frame: 6 weeks (from Baseline to end of Maintenance Period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Melperone HCl - 20 mg | Melperone HCl - 40 mg | Melperone HCl - 60 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 21 | 25
Scores on a scale | 0.7 (8.5) | 1.8 (12.9) | 0.9 (11.1) | 0.5 (6.4)
Statistical Analysis 1: Comparison: Melperone HCl - 20 mg vs Melperone HCl - 40 mg vs Melperone HCl - 60 mg vs Placebo; Only subjects with both a baseline and a post-baseline value are included; Test type: Superiority or Other; p = 0.9212, ANCOVA — Overall p-value using a one-way ANCOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: AEs were recorded from administration of study drug on Day 1 to 30 days after the last dose of study drug. SAEs were collected from when the informed consent and HIPAA (US sites only) were signed to 30 days after the last dose of study drug.
Description: All AEs, expected or unexpected, that occurred during the study, whether observed by the investigator or by the subject and whether or not these events were thought to be related to study drug, were reported and followed-up until resolved or until the investigator judged that further follow-up was not necessary.
Arm/Group | Melperone HCl - 20 mg | Melperone HCl - 40 mg | Melperone HCl - 60 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/15 | 2/19 | 2/25 | 0/30
Other Adverse Events (participants affected / at risk) | 6/15 | 8/19 | 10/25 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melperone HCl - 20 mg (N=15) | Melperone HCl - 40 mg (N=19) | Melperone HCl - 60 mg (N=25) | Placebo (N=30)
Parkinson's Disease (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Muscle strain (Investigations) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Melperone HCl - 20 mg (N=15) | Melperone HCl - 40 mg (N=19) | Melperone HCl - 60 mg (N=25) | Placebo (N=30)
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 1
Parkinson's Disease (Nervous system disorders) | 2 | 4 | 5 | 4
Somnolence (Nervous system disorders) | 2 | 3 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI could publish the results of the Study after the earlier of (a) the cooperative publication of the data, or (b) 18 months after Sponsor's final evaluation of all data; the PI will submit for review and approval any proposed abstracts and manuscripts at least 45 days prior to submission. The Institution and PI agree to delete any information the Sponsor deems confidential or proprietary; if the parties disagree, then they agree to meet prior to submission to discuss and resolve the issues.